CLINICAL TRIAL: NCT02038231
Title: Reducing Stress With Parenting-focused Mindfulness to Prevent Youth Substance Use
Brief Title: Parenting Mindfully Study
Acronym: PM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Inova Fairfax Hospital (Other)
Responsible Party: Principal Investigator, Tara M. Chaplin, Ph.D., Assistant Professor of Psychology, George Mason University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8753; R34DA034823 (NIH)
Record Dates: First submitted 2014-01-13; First posted 2014-01-16 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Substance Abuse; Risk Behaviors
Keywords: Adolescence; Substance abuse; Mindfulness
MeSH Terms: conditions — Substance-Related Disorders; Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parenting Mindfully Program (Experimental): Mindfulness program for parents of adolescents provided for 2 hours once per week for 8 weeks.
  Interventions: Behavioral: Parenting Mindfully Program
- Parent Education Program (Active Comparator): Group for parents of adolescents providing handouts and brief education to parents on topics of adolescence, family relations, and risk behaviors. Group meets 3 times over the course of 8 weeks for about 15 minutes per meeting.
  Interventions: Other: Parent Education Program

INTERVENTIONS:
Behavioral: Parenting Mindfully Program — see Arm Description.
  Arms: Parenting Mindfully Program
Other: Parent Education Program — See Arm Description.
  Arms: Parent Education Program

SUMMARY:
The goal of study is to develop and test a parenting-focused version of mindfulness intervention ("Parenting Mindfully") to reduce parent stress and prevent adolescent substance use and HIV risk behaviors (e.g., risky sex). The investigators hypothesize that Parenting Mindfully (PM) will decrease prevent adolescent substance use and HIV risk behaviors and intentions. Secondarily, PM will improve parenting, and decrease adolescent stress responses.

ELIGIBILITY:
Inclusion Criteria:

1. Family with a child between 12-16 years;
2. High parenting stress (mean score of >=3 on 2 questions adapted from the Perceived Stress Scale and the Parenting Stress Index).

Exclusion Criteria:

1. Diagnosis of mental retardation, autism or other pervasive developmental disorder for adolescent;
2. Current serious psychiatric or medical disorder (including current substance dependence) requiring immediate treatment for adolescent or parent- We will include those that are in treatment;
3. Medical condition that would preclude participation in gentle yoga (for parents)
4. Inadequate English proficiency to complete questionnaires for youth or parents.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2018-02 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change in Substance Use from pre-intervention through 12 months after the intervention | Pre-intervention, immediately post-intervention (8 weeks after the pre-intervention session), 6 months after the post-intervention session, and 12-month after the post-intervention session
  Measured by a combination of self-report on the Youth Risk Behavior Survey and a drug-use intentions questionnaire and urine toxicology and alcohol breathalyzer results.
Change in Adolescent Sex Behaviors from Pre-intervention Through 12 months following the intervention | Pre-intervention, immediately post-intervention (8 weeks after the pre-intervention session), 6 months after the post-intervention session, and 12-month after the post-intervention session
  Measured by self-report of onset of sex and risky sex behaviors on the Youth Risk Behavior Survey and a risky sexual behavior and intention questionnaire.

SECONDARY OUTCOMES:
Change in Parenting from Pre-Intervention to Post-Intervention | Pre-intervention, immediately post-intervention (8 weeks after the pre-intervention session)
  Measured by self-reported parenting behaviors on the Alabama Parenting Questionnaire and by parenting behaviors coded from videotapes of parent-adolescent interactions.
Change in Adolescent Stress Responses from Pre-Intervention to Post-Intervention | Pre-intervention, immediately post-intervention (8 weeks after the pre-intervention session)
  Measured by adolescent's reported emotions, observed emotion expressions, and heart rate, blood pressure, and cortisol levels in response to stressful parent-adolescent interactions.

CONTACTS AND LOCATIONS:
Locations (1):
- George Mason University Department of Psychology, Fairfax, Virginia, United States

REFERENCES:
- [Derived] Chaplin TM, Mauro KL, Curby TW, Niehaus C, Fischer S, Turpyn CC, Martelli AM, Miller AB, Leichtweis RN, Baer R, Sinha R. Effects of A Parenting-Focused Mindfulness Intervention on Adolescent Substance Use and Psychopathology: A Randomized Controlled Trial. Res Child Adolesc Psychopathol. 2021 Jul;49(7):861-875. doi: 10.1007/s10802-021-00782-4. Epub 2021 Feb 23. PMID 33620662